CLINICAL TRIAL: NCT03589209
Title: Preoperative CT Scan Analysis to Predict Perioperative Round Window Visibility Through the Posterior Tympanotoy in Cochlear Implant Surgery
Brief Title: Prediciton of the Round Window Visibility Through Posterior Tympanotomy by CT Scan Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7052
Record Dates: First submitted 2018-07-04; First posted 2018-07-17 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-06

CONDITIONS: Tympanostomy Tube Insertion
Keywords: Round window visibility; Cochlear implantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is difficult to predict the intraoperative visibility of the round window through the posterior Tympanostomy. In case of non-visualization, the surgeon may have to change operative technique during cochlear implant surgery.

The primary purpose of the study is to define relevant CT measurements on the preoperative scanner to predict the perioperative visibility of the round window. Define relevant CT measurements on the preoperative scanner to predict the perioperative visibility of the round window.

The secondary purpose is to validate the investigator's scanner reading protocol for a prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Aged subject from 9 months and over
* Implanted cochlear subject in the ENT department of Strasbourg between 1st January 2010 and 1st March 2018
* Subject (or the holders of parental authority in the case of minors) having agreed to the use of medical data for the purpose of this research.

Exclusion Criteria:

* Refusal of the patient to participate in the study
* CROP does not make it possible to evaluate the visibility of the FR
* Preoperative or uninterpretable scanner
* Major anatomical malformation
* Subject under the protection of justice
* Subject under guardianship or curatorship

Min Age: 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Implanted cochlear subject in the ENT department of Strasbourg between 1st January 2010 and 1st March 2018
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Measure of the correlation between preoperative CT measurements and the visibility of the round window observed intraoperatively (based on the operative records) | 1 day after cochlear implantation surgery
  Analysis of patient records (operative reports and preoperative CT-scan) from patients who underwent cochlear implantation between 01/01/2010 and 01/03/2018.

CONTACTS AND LOCATIONS:
Overall Officials: Anne CHARPIOT, MD, PhD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service D'Orl Et de Chirurgie Cervico-Faciale, Strasbourg, France